CLINICAL TRIAL: NCT00538031
Title: Randomized Pilot Trial of Oral Cyclophosphamide Versus Oral Cyclophosphamide With Celecoxib for Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Cyclophosphamide With or Without Celecoxib in Treating Patients With Recurrent or Persistent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03092; NCI-2009-01597 (Registry Identifier: NCI CTRP); CDR0000567043 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Fallopian Tube Cancer; Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cyclophosphamide; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive oral cyclophosphamide once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide
- Arm II (Experimental): Patients receive oral cyclophosphamide once daily and oral celecoxib twice daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: celecoxib

INTERVENTIONS:
Drug: cyclophosphamide — Given orally
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Drug: celecoxib — Given orally
  Other Names: Celebrex; SC-58635; YM 177
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cyclophosphamide together with celecoxib may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving cyclophosphamide together with celecoxib works compared to cyclophosphamide alone in treating patients with recurrent or persistent ovarian epithelial, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess the response rates in patients with recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal cancer who are treated with oral cyclophosphamide alone or oral cyclophosphamide with celecoxib.

II. To assess the time to disease progression in this group of patients. III. To further describe the toxicities of oral cyclophosphamide with or without celecoxib in the above patient population.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral cyclophosphamide once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive oral cyclophosphamide once daily and oral celecoxib twice daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion

* Patients with recurrent or residual epithelial ovarian, Fallopian tube, or primary papillary peritoneal cancer, which has been histologically confirmed regardless of prior treatment
* Patients with measurable disease or rising CA-125 to levels at least twice normal (the CA-125 increase must be documented by two independent measurements at least 4 weeks apart)
* Patient must have adequate renal function documented by a creatinine < 1.5
* Patients must have adequate bone marrow function as evidenced by an absolute neutrophil count of > 1.5 x 10^9/L and a platelet count > 100 x 10^9/L
* Patients must have a Karnofsky performance status of 60-100%
* Patient must be capable of understanding the nature of the trial and must give written informed consent
* Patients must have life expectancy of at least three months
* Patients with brain metastases which at the time of study enrollment are controlled and do not require treatment with corticosteroids are eligible

Exclusion

* Patients who have had radiotherapy or chemotherapy within three weeks prior to anticipated first day of dosing (patients must be fully recovered from the acute effects of any prior chemotherapy or radiotherapy
* Patient with unstable or severe intercurrent medical conditions or active, uncontrolled infection
* Patients with history of bleeding peptic ulcer within last 3 months
* Patients undergoing therapy with other investigational agents (patients must have recovered from all acute effects of previously administered investigational agents and sufficient time must have elapsed since last administration to ensure the drug interactions not occur during this study
* Patients who are allergic to sulfa drugs
* Pregnant women will be excluded from this study due to the potential of harm to the fetus
* Patients with clinically significant cardiovascular disease (e.g. uncontrolled hypertension, myocardial infarction unstable angina), New York heart association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or grade II or greater peripheral vascular disease within 1 year prior to study entry
* Subjects with hypertension are eligible if their blood pressure as been normal while on a stable dose of medication for at least one year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-12-22 (Actual); Primary Completion 2011-04-21 (Actual); Study Completion 2019-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - City of Hope Medical Group Inc, Pasadena, California

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31279962/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Cyclophosphamide Alone): Patients receive 50 mg oral cyclophosphamide once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
- Arm II (Cyclophosphamide + Celecoxib): Patients receive 50 mg oral cyclophosphamide once daily and 400 mg oral celecoxib twice daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Cyclophosphamide Alone) | Arm II (Cyclophosphamide + Celecoxib)
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cyclophosphamide Alone) | Arm II (Cyclophosphamide + Celecoxib) | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Median (Full Range); unit: years] | 60 [27 to 79] | 61 [48 to 80] | 61 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 5 | 9
  Hispanic | 1 | 5 | 6
  White non-Hispanic | 20 | 15 | 35
  Native American | 1 | 0 | 1
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52
Karnofsky performance status [Median (Full Range); unit: units on a scale] — 100 Normal no complaints; no evidence of disease 90 Normal activity; minor signs\symptoms of disease 80 Normal activity with effort; some signs\symptoms of disease 70 Cares for self; unable to carry on normal activity or to do active work 60 Requires occasional assistance, can care for most personal needs 50 Requires considerable assistance and frequent medical care 40 Disabled; requires special care\assistance 30 Severely disabled; hospital admission is indicated, death not imminent 20 Very sick; hospital admission necessary; active supportive treatment 10 Moribund 0 Dead
  units on a scale | 90 [70 to 100] | 90 [60 to 100] | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cyclophosphamide Alone) | Arm II (Cyclophosphamide + Celecoxib)
Number analyzed (Participants) | 26 | 26
Participants | 1 | 1

2. Primary Outcome: Time to Treatment Failure
Description: Estimated using the product-limit method of Kaplan and Meier. Time to treatment failure is defined as the time from initial treatment to discontinuation of treatment for any reason, including progression of disease, treatment toxicity, and death.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Cyclophosphamide Alone) | Arm II (Cyclophosphamide + Celecoxib)
Number analyzed (Participants) | 26 | 26
Months | 1.84 [1.68 to 2.76] | 1.92 [1.64 to 5.22]
Statistical Analysis 1: Comparison: Arm I (Cyclophosphamide Alone) vs Arm II (Cyclophosphamide + Celecoxib); Test type: Other; p = 0.61, Log Rank

3. Primary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier. From time of initial treatment to death from any cause.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Cyclophosphamide Alone) | Arm II (Cyclophosphamide + Celecoxib)
Number analyzed (Participants) | 26 | 26
Months | 9.69 [3.84 to 13.18] | 12.55 [6.67 to 17.61]
Statistical Analysis 1: Comparison: Arm I (Cyclophosphamide Alone) vs Arm II (Cyclophosphamide + Celecoxib); Test type: Other; p = 0.95, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 7 years and 3 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm I (Cyclophosphamide Alone) | Arm II (Cyclophosphamide + Celecoxib)
All-Cause Mortality (participants affected / at risk) | 26/26 | 26/26
Serious Adverse Events (participants affected / at risk) | 4/26 | 8/26
Other Adverse Events (participants affected / at risk) | 26/26 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cyclophosphamide Alone) (N=26) | Arm II (Cyclophosphamide + Celecoxib) (N=26)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 0 (0) | 2 (2)
General symptom (General disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cyclophosphamide Alone) (N=26) | Arm II (Cyclophosphamide + Celecoxib) (N=26)
Dyspareunia (General disorders) | 0 (0) | 1 (1)
Haemorrhage NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 13 (32) | 17 (41)
Lymphangiopathy NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (4) | 3 (9)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 4 (4)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 15 (22) | 15 (36)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 7 (11) | 10 (16)
Diarrhea (Gastrointestinal disorders) | 11 (17) | 11 (21)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 5 (8)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 4 (6)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (21) | 14 (26)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (9) | 10 (13)
Chest pain (General disorders) | 4 (5) | 2 (2)
Chills (General disorders) | 2 (2) | 4 (4)
Edema (General disorders) | 0 (0) | 2 (3)
Edema limbs (General disorders) | 3 (4) | 3 (4)
Fatigue (General disorders) | 13 (27) | 16 (39)
Fever (General disorders) | 2 (2) | 4 (5)
General symptom (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Oedema NOS (General disorders) | 0 (0) | 2 (4)
Pain (General disorders) | 10 (14) | 13 (46)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (9) | 9 (14)
Alkaline phosphatase increased (Investigations) | 15 (31) | 9 (14)
Aspartate aminotransferase increased (Investigations) | 19 (34) | 17 (40)
Bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (4) | 5 (15)
Leukocyte count decreased (Investigations) | 8 (22) | 6 (11)
Leukopenia (Investigations) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (5) | 5 (6)
Lymphopenia (Investigations) | 4 (5) | 3 (10)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (6)
Platelet count decreased (Investigations) | 2 (4) | 2 (2)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 8 (9) | 9 (14)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (3) | 3 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (16) | 4 (5)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 5 (10)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 3 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (9) | 6 (13)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (3) | 2 (4)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (4) | 8 (17)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 8 (12) | 6 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 4 (11)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 7 (8) | 3 (6)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (2) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (9) | 6 (10)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Taste alteration (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (11) | 8 (10)
Depression (Psychiatric disorders) | 5 (7) | 2 (7)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 2 (2)
Blood urine present (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (3)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 3 (5)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 2 (6) | 5 (10)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 3 (11)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 9 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT00538031/Prot_SAP_000.pdf